CLINICAL TRIAL: NCT06083571
Title: Efficacy of Nasal Migraine Cocktail Used In Pediatric Emergency Department: A Clinical Trial
Brief Title: Intranasal Ketorolac Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The eligibility criteria within the protocol led to the exclusion of a large proportion of potential participants, thereby limiting enrollment. During the conceptualization phase, the number of eligible patients was overestimated.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Assertio Holdings, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202307050
Record Dates: First submitted 2023-09-18; First posted 2023-10-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Ketorolac; Prochlorperazine; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Patients (Experimental): Intranasal ketorolac (1 spray (15.75mg) if 15kg-29.9kg and 2 sprays (31.5mg) if 30kg or heavier and oral adjuncts oral Prochlorperazine (Between 15-25 kg: dose of 2.5 mg; 26-50 kg: dose of 5 mg; > 50 kg: dose of 10 mg, single maximum dose 10 mg) and oral Diphenhydramine (Between 15-25 kg: dose of 12.5 mg; 26-50 kg: dose of 25 mg; > 50 kg: dose of 50 mg, single maximum dose 50mg)
  Interventions: Drug: Ketorolac; Drug: Prochlorperazine; Drug: Diphenhydramine
- Intravenous Patients (Active Comparator): IV ketorolac (0.5 mg/kg, maximum single dose of 30 mg) with oral adjuncts oral Prochlorperazine (Between 15-25 kg: dose of 2.5 mg; 26-50 kg: dose of 5 mg; > 50 kg: dose of 10 mg, single maximum dose 10 mg) and oral Diphenhydramine (Between 15-25 kg: dose of 12.5 mg; 26-50 kg: dose of 25 mg; > 50 kg: dose of 50 mg, single maximum dose 50mg)
  Interventions: Drug: Ketorolac; Drug: Prochlorperazine; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Ketorolac — Non-inferiority
  Other Names: Sprix
Drug: Prochlorperazine — Adjunct
  Other Names: Compazine
Drug: Diphenhydramine — Adjunct
  Other Names: Benadryl

SUMMARY:
The purpose of this study is to determine if intranasal (IN) Ketorolac in combination with oral Prochlorperazine and Diphenhydramine is non-inferior to current migraine management which involves use of intravenous (IV) Ketorolac and oral adjuncts Prochlorperazine and diphenhydramine for reducing pain intensity in children with migraine headaches.

The investigators hypothesize that IN ketorolac combined with these oral adjuncts is non-inferior to IV ketorolac and oral adjuncts in reducing acute migraine headache pain by a minimum clinically significant difference within 60 minutes of administration.

ELIGIBILITY:
Inclusion Criteria:

* A headache that fulfills at least three of the six following criteria: i) moderate to severe episode of impaired daily activities; ii) focal localization of headache (focal meaning unilateral, bifrontal, bitemporal, or biparietal); iii) pulsatile description; iv) nausea or vomiting or abdominal pain; v) photophobia or phonophobia or avoidance of light and noise; and vi) symptoms increasing with activity or resolving by rest
* Pain 4/10 on the validated Faces Pain Scale
* Headache duration between 1 and 72 hours

Exclusion Criteria:

* Any contraindication to receiving ketorolac (e.g. known allergy, known peptic ulcer disease, gastrointestinal bleeding, hepatic impairment (patients with known aspartate aminotransferase (AST) > 60 units/L "OR" alanine aminotransferase (ALT) > 40 units/L "OR" total bilirubin > 1.2 mg/dl)
* Renal impairment (patients with known estimated glomerular filtration rate of < 90 mL/min/1.73m2)
* Known bleeding disorders
* Receipt of an NSAID (e.g. ibuprofen, naproxen, naproxen/sumatriptan) within previous six hours
* Receipt of oral prochlorperazine or metoclopramide or diphenhydramine within 12 hours prior to presentation
* Presence of intranasal obstruction (e.g. mucous or blood) that cannot be readily cleared using suction or nose blowing
* Inability to speak English
* Patients with a concurrent diagnosis of traumatic brain injury
* Unable to complete self-report measures of pain or questionnaires (e.g. developmental delay, neurologic impairment)
* Critical illness
* Frequent use of drugs for headache (defined as regular intake of analgesics for acute headaches on more than 10 days per month)
* Patients refusing to take oral adjuncts or unable to tolerate oral medications will be excluded from the trial.
* Patients currently on the following medications will also be excluded from the study as there are contraindications for use of Ketorolac with use of these medications: antiplatelets (i.e. salicylates, aspirin, clopidogrel, ticagrelor), Anticoagulants (i.e. warfarin, rivaroxaban, apixaban, dabigatran, enoxaparin, and heparin), angiotensin-converting enzyme inhibitors/angiotensin receptor blockers (losartan, Lisinopril), cyclosporine or tacrolimus, furosemide, bumetanide, spironolactone, hydrochlorothiazide, digoxin, lithium, methotrexate, probenecid, some selective serotonin reuptake inhibitors (including i.e. citalopram, escitalopram, sertraline), antipsychotics (i.e. Quetiapine, risperidone, aripiprazole, haloperidol), tranylcypromine, oxybates, oral potassium citrate, and Anticholinergics (i.e. amantadine).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on the 10 point Faces Pain Scale-Revised in 2 hours | Baseline (within 15 minutes prior to receiving the study drug or as close to this time frame as possible) and then at 10 minutes, 30 minutes, 60 minutes, and 120 minutes (or as close to this time frame as possible)
  The Faces Pain Scale - Revised. This is a 10-point pain scale (0-10) that has been validated for the use in children greater than 4 years of age in the ED; is one of the self-report measures of pain recommended for research in children; and is commonly used as the primary outcome in Emergency Department research. Lower numbers are better outcomes.

SECONDARY OUTCOMES:
Response Rate- 2/10 score difference of pain on the Faces Pain Scale- Revised | 10 minutes after medication given
  Response rate is defined as the number of participants with a pain scale change of at least 2/10 on The Faces Pain Scale - Revised from baseline to 10 minutes after medication given. The Faces Pain Scale - Revised. The Faces Pain Scale - Revised is a 10-point pain scale that has been validated for the use in children greater than 4 years of age in the Emergency Department; is one of the self-report measures of pain recommended for research in children; and is commonly used as the primary outcome in Emergency Department research. The lower numbers on this scale report better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Rifkin, MD, Principal Investigator — Washington University in St. Louis: st. louis childrens hospital
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuensting LL, DeBoer S, Holleran R, Shultz BL, Steinmann RA, Venella J. Difficult venous access in children: taking control. J Emerg Nurs. 2009 Sep;35(5):419-24. doi: 10.1016/j.jen.2009.01.014. Epub 2009 Mar 21. No abstract available. PMID 19748021
- [Background] Tsze DS, Lubell TR, Carter RC, Chernick LS, DePeter KC, McLaren SH, Kwok MY, Roskind CG, Gonzalez AE, Fan W, Babineau SE, Friedman BW, Dayan PS. Intranasal ketorolac versus intravenous ketorolac for treatment of migraine headaches in children: A randomized clinical trial. Acad Emerg Med. 2022 Apr;29(4):465-475. doi: 10.1111/acem.14422. Epub 2021 Dec 13. PMID 34822214